CLINICAL TRIAL: NCT01594437
Title: Phase 1 Study of TCN-202 (Human Anti-Cytomegalovirus Monoclonal Antibody) in Healthy Adult Volunteers
Brief Title: Safety Study of Human Anti-Cytomegalovirus Monoclonal Antibody
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theraclone Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCN-202-001
Record Dates: First submitted 2012-05-05; First posted 2012-05-09 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus; Monoclonal antibody
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCN-202 (Experimental)
  Interventions: Biological: TCN-202
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TCN-202 — Human monoclonal neutralizing antibody that recognizes a broadly conserved functional epitope on HCMV. One or two doses will be administered by intravenous infusion.
  Other Names: Human Anti-Cytomegalovirus Monoclonal Antibody
  Arms: TCN-202
Biological: Placebo — One or two doses administered by intravenous infusion.
  Other Names: 0.9% Sodium chloride for Injection, USP
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety profile in healthy adult volunteers of single or multiple intravenous administrations of TCN-202 as compared with placebo.

DETAILED DESCRIPTION:
Human cytomegalovirus (HCMV) disease remains an unmet medical need: In the US, the estimated prevalence of congenital HCMV infection is ~1% and is one of the leading causes of permanent hearing loss and neurological deficits in children. In immunocompromised individuals such as transplant recipients it can cause serious life-threatening disease and may significantly increase the risk of graft rejection. As existing therapies for HCMV can have serious side effects, there remains a medical need for safe and effective treatment of HCMV disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* Normal lab tests

Exclusion Criteria:

* Prior treatment with monoclonal antibody

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events | 60 days post infusion
  Adverse events will be determined by physical examinations, vital signs, serial electrocardiograms, and clinical laboratory abnormalities (hematology, chemistry, and urinalysis).

SECONDARY OUTCOMES:
Peak serum concentration (Cmax) of TCN-202 | 1 day post infusion
Number of subjects who develop anti-TCN-202 anti-drug antibodies (immunogenicity) | 60 days post infusion
  Immunogenicity will be assessed based on induction of TCN-202 anti-drug antibodies.
Area under the concentration time curve (AUC) of TCN-202 | 60 days post infusion
Time to maximum serum concentration (Tmax) of TCN-202 | 1 day post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, FACP, Principal Investigator — SNBL Clinical Pharmacology Center
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States